CLINICAL TRIAL: NCT02968654
Title: Transfusion Strategies in Acute Brain Injured Patients. A Prospective Multicenter Randomized Study.
Brief Title: TRansfusion Strategies in Acute Brain INjured Patients
Acronym: TRAIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erasme University Hospital (Other)
Collaborators: European Society of Intensive Care Medicine (Other)
Responsible Party: Principal Investigator, Fabio Taccone, Professor, Erasme University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P2015/327; NCT02962349 (obsolete NCT alias)
Record Dates: First submitted 2016-11-11; First posted 2016-11-18 (Estimated); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Acute Brain Injury; Blood Transfusion
Keywords: Blood Transfusion; Brain Injury; Outcome; Hemoglobin
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Restrictive Transfusion Strategy (Other): "Blood Transfusion" will be given when hemoglobin concentration will be below 7 g/dL (as suggested by current guidelines in "general" ICU population)
  Interventions: Procedure: Restrictive Transfusion Strategy
- Liberal Transfusion Strategy (Other): "Blood Transfusion" will be given when hemoglobin concentration will be below 9 g/dL
  Interventions: Procedure: Liberal Transfusion Strategy

INTERVENTIONS:
Procedure: Restrictive Transfusion Strategy — Patients will be randomized when hemoglobin levels will be below 9 g/dl. Patients randomized to the "Restrictive Transfusion Strategy" will receive blood transfusion whenever their Hb concentration is < 7 g/dl. All patients should preferably receive one unit of blood transfusion at a time. The duration of the intervention is 28 days after randomization or until hospital discharge. Daily assessment of hemoglobin levels are mandatory only during the ICU stay. No other procedures and or interventions are scheduled. General management of patients will be conducted according to international guidelines; however, local protocols and procedures are allowed.
  Arms: Restrictive Transfusion Strategy
Procedure: Liberal Transfusion Strategy — Patients will be randomized when hemoglobin levels will be below 9 g/dl. Patients randomized to the "Liberal Transfusion Strategy" will receive blood transfusion whenever their Hb concentration is < 7 g/dl. All patients should preferably receive one unit of blood transfusion at a time. The duration of the intervention is 28 days after randomization or until hospital discharge. Daily assessment of hemoglobin levels are mandatory only during the ICU stay. No other procedures and or interventions are scheduled. General management of patients will be conducted according to international guidelines; however, local protocols and procedures are allowed.
  Arms: Liberal Transfusion Strategy

SUMMARY:
To compare a "liberal" and a "restrictive" strategy to administer blood transfusions in critically ill patients with a primary brain injury.

DETAILED DESCRIPTION:
Although blood transfusions can be lifesaving in severe hemorrhage, they can also have potential complications. As anemia has also been associated with poor outcomes in critically ill patients, determining an optimal transfusion trigger is a real challenge for clinicians. This is even more important in patients with acute brain injury who were not specifically evaluated in previous large randomized clinical trials dealing with the optimal transfusion threshold. Neurological patients may be particularly sensitive to anemic brain hypoxia because of the exhausted cerebrovascular reserve, which adjusts cerebral blood flow to tissue oxygen demand.

This prospective, multicenter, randomized, pragmatic trial will compare two different strategies for red blood cell transfusion in patients with acute brain injury: a "liberal" strategy in which the aim is to maintain hemoglobin (Hb) concentrations greater than 9 g/dL and a "restrictive" approach in which the aim is to maintain Hb concentrations greater than 7 g/dL. The target population is patients suffering from traumatic brain injury (TBI), subarachnoid hemorrhage (SAH) or intracranial hemorrhage (ICH).

The primary outcome is neurological outcome, evaluated using the extended Glasgow Outcome Scale (eGOS), at 180 days after the initial injury. Secondary outcomes include, amongst others, 28-day survival, intensive care unit (ICU) and hospital lengths of stay, the occurrence of extra-cerebral organ dysfunction/failure and the development of any infection or thromboembolic events (venous or arterial).

The estimated sample size is 794 patients to demonstrate a reduction in the primary outcome (i.e. unfavorable neurological outcome) from 50% to 30% between groups (397 patients in each arm). The study will be initiated in September 2016 in several European ICUs and is expected at least 6 years.

The results of this trial will help to improve blood product and transfusion use in this specific patient population and will provide additional data in some sub-groups of patients at high-risk of brain ischemia, such as those with intracranial hypertension or cerebral vasospasm.

ELIGIBILITY:
Inclusion Criteria:

* Glasgow Coma Score (GCS) ≤ 13 on randomization
* Expected ICU stay > 72 hours
* hemoglobin (Hb) concentration ≤ 9 g/dL within 10 days from brain injury

Exclusion Criteria:

1. Post-anoxic coma; status epilepticus without underlying brain injury; central nervous system (CNS) infections (community-acquired; hospital-acquired; ventriculitis; post-operative)
2. Known previous neurological disease, causing significant cognitive and/or motor handicap
3. ICH due to arterio-venous malformation (AVM) or brain tumor
4. Inability (religious reasons) or reduced ability (lack of compatible blood) to receive blood products
5. Active and uncontrolled bleeding at the time of enrollment
6. GCS of 3 with both pupils fixed and dilated; brain death or imminent death (within 24 hours)
7. Pregnancy
8. Medical need to correct anemia (e.g., active coronary disease or severe cardiac disease) with target Hb levels > 9 g/dL
9. do-not-escalate (DNE) orders
10. Previous allo-immunization due to transfusion, limiting red blood cells (RBC) availability

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 850 (Actual)
Dates: Start 2016-09-13 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Unfavorable Neurological Outcome | 180 days after randomization
  Unfavorable neurological outcome is defined by the extended Glasgow Outcome Scale (eGOS) of 1-5

SECONDARY OUTCOMES:
Survival | 28 days
  28 days Survival
Changes in the Glasgow Coma Score (GCS) over time | 28 days
  modification of GCS from admission over the first week and vs. the last available
ICU length of stay | 180 days
  length of ICU stay
Hospital length of stay | 180 days
  length oh hospital stay
Presence and severity of extra-cerebral organ dysfunction/failure | 28 days
  Daily sequential organ failure assessment (SOFA) score
Infection rate | 28 days
  Occurrence of any infection over the first 28 days after randomization
Composite outcome | 28 days
  Death and Organ Failure (defined as at least one extra-cerebral organ failure, according to the specific SOFA sub-score > 2)
Brain Oxygen Pressure | 28 days
  Absolute values of brain oxygen pressure (PbO2) for those patients where this neuromonitoring has been implemented, according to the decision of the attending physician
Daily Fluid Balance | 28 days
  Assessment of the daily fluid balance
Serious Adverse Events (SAE) | 28 days
  Any of the "SAE" as described in the study protocol

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Erasme, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Taleb C, Gouvea Bogossian E, Bittencour Rynkowski C, Moller K, Lormans P, Quintana Diaz M, Caricato A, Zattera L, Kurtz P, Meyfroidt G, Quintard H, Dias MC, Giacomucci A, Castelain C, Chabanne R, Marcos-Neira P, Bendel S, Alsheikhly AS, Elbahnasawy M, Gay S, D'Onofrio M, Popugaev KA, Markou N, Bouzat P, Vincent JL, Taccone FS; TRAIN Study Trial Group. Liberal versus restrictive transfusion strategies in subarachnoid hemorrhage: a secondary analysis of the TRAIN study. Crit Care. 2025 Feb 7;29(1):67. doi: 10.1186/s13054-025-05270-5. PMID 39920710
- [Derived] Taccone FS, Rynkowski CB, Moller K, Lormans P, Quintana-Diaz M, Caricato A, Cardoso Ferreira MA, Badenes R, Kurtz P, Sondergaard CB, Colpaert K, Petterson L, Quintard H, Cinotti R, Gouvea Bogossian E, Righy C, Silva S, Roman-Pognuz E, Vandewaeter C, Lemke D, Huet O, Mahmoodpoor A, Blandino Ortiz A, van der Jagt M, Chabanne R, Videtta W, Bouzat P, Vincent JL; TRAIN Study Group. Restrictive vs Liberal Transfusion Strategy in Patients With Acute Brain Injury: The TRAIN Randomized Clinical Trial. JAMA. 2024 Nov 19;332(19):1623-1633. doi: 10.1001/jama.2024.20424. PMID 39382241
- [Derived] Taccone FS, Badenes R, Rynkowski CB, Bouzat P, Caricato A, Kurtz P, Moller K, Diaz MQ, Van Der Jagt M, Videtta W, Vincent JL. TRansfusion strategies in Acute brain INjured patients (TRAIN): a prospective multicenter randomized interventional trial protocol. Trials. 2023 Jan 7;24(1):20. doi: 10.1186/s13063-022-07061-7. PMID 36611210